CLINICAL TRIAL: NCT02144467
Title: The Establishment of Large-sample Database of "Multiple-MRI/Gene/Cognition"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Yu-Feng ZANG, deputy director, Hangzhou Normal University
Other Study IDs: HNU_CCBD_LargeSampleCollection
Record Dates: First submitted 2014-05-14; First posted 2014-05-22 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Multiple-MRI, Gene, Cognition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral Venous Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Large-sample healthy participants: MRI scanning.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — fMRI, sMRI, ASL and DTI

SUMMARY:
Aim to establish a large-sample database of "Multiple-MRI/Gene/Cognition" for healthy Chinese (sample number, 5000; age, 6-70 years). This is a fundamental but very necessary work for future researches such as development, aging, relation of gene and behavior, relation of gene and neuroimaging, relation of behavior and neuroimaging. Importantly, this work will provide a norm for researches on psychological or neurological patients. This large-sample will be shared with world-wide researchers.

DETAILED DESCRIPTION:
A part of data have been used in a publication which is preparing to submit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese
* Age: 6-70 years old
* Right handed
* No smoking or alcoholic addiction

Exclusion Criteria:

* Psychological or neurological patients
* Hypertension or cardiopathy patients
* Pregnant woman
* Take medicine or drink tea/coffee before scanning-

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Hangzhou, China.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-05-08 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Estimated)

PRIMARY OUTCOMES:
The distribution of the amplitude of blood oxygenation level dependent(BOLD) signal in healthy subjects | up to 15 months
  The amplitude of BOLD-functional magnetic resonance imaging(fMRI) signal is a common measure to estimate the brain activity during resting-state. We try to establish its distribution on healthy subjects, which could be a control to examine abnormal brain function in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Feng ZANG, M.D., Principal Investigator — Hangzhou Normal University, Center for Cognition and Brain Disorder
Locations (1):
- Hangzhou Normal University,Center for Cognition and Brain Disorder, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The data cannot be share with other researchers right now. It will be shared two years later.

REFERENCES:
- [Derived] Jing Y, Zhao N, Deng XP, Feng ZJ, Huang GF, Meng M, Zang YF, Wang J. Pregenual or subgenual anterior cingulate cortex as potential effective region for brain stimulation of depression. Brain Behav. 2020 Apr;10(4):e01591. doi: 10.1002/brb3.1591. Epub 2020 Mar 8. PMID 32147973